CLINICAL TRIAL: NCT07322523
Title: Validation of Smartwatch Technology for Preoperative Monitoring of Sleep Quality, Anxiety, and Vital Signs in Patients Undergoing Disc Herniation Surgery
Brief Title: Smartwatch Accuracy for Measuring Vitals and Anxiety Before Disc Surgery
Status: Recruiting | Type: Observational
Sponsor: Halil Kalaycı (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Sponsor-Investigator, Halil Kalaycı, Res. Asst., TC Erciyes University
Organization: TC Erciyes University (Other)
Other Study IDs: 96681246
Record Dates: First submitted 2025-12-08; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Disc Herniations; Disc Herniation, Lumbar; Cervical Disc Herniation; Preoperative Anxiety Score; Sleep Quality; Preoperative Care; Vital Signs Monitoring; Smart Watch; Wearable Devices; Surgical Nursing
Keywords: Disc herniations; wearable devices; smart watch; vital signs monitoring; sleep quality; anxiety; surgical nursing,; preoperative
MeSH Terms: conditions — Intervertebral Disc Displacement; Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preoperative Disc Herniation Patients: This group consists of hospitalized adult patients scheduled for intervertebral disc herniation surgery whose preliminary examinations are complete. Measurements will be taken at two different time points: the night before surgery and the morning of the surgery. Patients' vital signs (blood pressure, pulse, oxygen saturation) will be determined using standard medical devices, while anxiety and sleep quality will be determined via validated clinical scales. All these values will be collected simultaneously using smartwatches (Samsung).

SUMMARY:
This study aims to verify the accuracy of blood pressure, heart rate, blood oxygen saturation, anxiety level, and sleep cycle data measurements obtained from Samsung smartwatches compared to the currently accepted method used in patients with disc herniation undergoing the preoperative period.

ELIGIBILITY:
Inclusion Criteria:

* 22 years and older
* Currently receiving preoperative care/assessment for disc herniation surgery.
* No history of any cardiovascular disease other than controlled hypertension.
* Willingness to wear the smartwatch for a minimum of 8 consecutive hours during the night before surgery.
* Ability to follow all instructions related to the smartwatch operation and data collection independently.
* No known allergy to nickel.

Exclusion Criteria:

* Patients who are currently receiving prescribed medication specifically for sleep in the clinical setting.
* Refusal or unwillingness to participate in the study.
* The participant fails to wear the smartwatch correctly or appropriately as per study instructions, leading to incomplete or unreliable data collection.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises adult inpatients admitted to the Neurosurgical Ward of the university hospital due to intervertebral disc herniation for preoperative assessment and monitoring.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure (BP) (Medical-Grade) | Evening before surgery; Morning before surgery.
  One measurement will be taken from both the patient's right and left arm using a calibrated medical-grade sphygmomanometer (BP cuff) at each time point. Both systolic and diastolic pressure will be recorded separately.
Heart Rate (HR) (Medical-Grade) | Evening before surgery; Morning before surgery.
  HR will be taken using a finger pulse oximeter on the finger of the same arm as the smartwatch at each time point.
Blood Oxygen Saturation (SpO2) (Medical-Grade) | Evening before surgery; Morning before surgery.
  SpO2 will be taken using a finger pulse oximeter on the finger of the same arm as the smartwatch at each time point.
State-Trait Anxiety Inventory (STAI) Score | Evening before surgery; Morning before surgery.
  The evening before surgery: Both the State-Trait Anxiety Inventory (STAI) State and Trait anxiety scores will be recorded. The morning before surgery: Only the State Anxiety Inventory score will be recorded. Both the State and Trait forms of the STAI include reverse-scored items. Total scores are calculated for each form, with higher scores reflecting higher levels of anxiety.
Richards-Campbell Sleep Questionnaire (RCSQ) Score | Evening before surgery; Morning before surgery
  Sleep quality will be measured twice using the Richards-Campbell Sleep Questionnaire (RCSQ): 1) The evening before surgery, to assess the night immediately before the decision to operate. 2) The morning before surgery, assess the preoperative night spent in the hospital. The total score is calculated using the first five items of the scale, with the noise item excluded from scoring. Scores of 0-25 indicate very poor sleep, while scores of 76-100 indicate very good sleep.
Blood Pressure (BP) (Measured via Wrist) | Evening before surgery; Morning before surgery.
  Blood pressure will be measured using a smartwatch twice: once on the evening before surgery and once on the morning of surgery. On both occasions, the smartwatch-based measurement will be obtained immediately prior to the medical blood pressure measurement. All measurements will be obtained from the same preoperatively designated wrist without changing sides. Systolic and diastolic blood pressure values obtained from the smartwatch will be recorded separately.
Heart Rate (HR) (Measured via Wrist) | Evening before surgery; Morning before surgery.
  Heart rate (HR) will be measured at the wrist using a smartwatch. During measurement, a simultaneous reference reading will be obtained from the finger of the same arm using a finger pulse oximeter, with the time interval between devices kept to a minimum.
Blood Oxygen Saturation (SpO2) (Measured via Wrist) | Evening before surgery; Morning before surgery.
  Peripheral oxygen saturation (SpO₂) will be measured at the wrist using a smartwatch. During measurement, a simultaneous reference reading will be obtained from the finger of the same arm using a finger pulse oximeter, with the time interval between devices kept to a minimum.
Anxiety Metric (Measured via Wrist) | Evening before surgery; Morning before surgery.
  Anxiety level will be assessed using a smartwatch. The smartwatch categorizes anxiety into four levels: relaxed, low, moderate, and high. To minimize the potential influence of self-awareness of questionnaire results, the smartwatch-based assessment will be conducted after completion of the STAI.
Sleep Quality (Measured via Wrist) | Single report obtained from continuous monitoring during the entire Night Before Surgery (from the evening when the watch is put on until the morning).
  Sleep will be continuously monitored using a smartwatch throughout the preoperative night. At the end of the monitoring period, sleep quality will be quantified using a score ranging from 0 to 100, with higher scores reflecting better sleep quality.
Sleep Duration (Measured via Wrist) | Single report obtained from continuous monitoring during the entire Night Before Surgery (from the evening when the watch is put on until the morning).
  Sleep duration will be continuously monitored using a smartwatch throughout the night. Total sleep duration will be reported in hours and minutes. In addition to total sleep duration, time spent in light sleep, REM sleep, wakefulness, and deep sleep will be reported as subcomponents. All sleep-related durations will be recorded separately in hours and minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
SPSS data